CLINICAL TRIAL: NCT07378384
Title: Effect of Virtual Simulation Games on Nursing Students' Knowledge, Skills, Confidence and Satisfaction in CVC Care
Brief Title: The Effect of Virtual Simulation Games on Nursing Students' Knowledge, Skills, Confidence and Satisfaction in CVC Care
Acronym: CVC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kandemir özsoy (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Zeynep Kandemir özsoy, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IKCU-NURSING-VIRTUALSIM-CVC-20
Record Dates: First submitted 2026-01-20; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Nurse Education
Keywords: Virtual Simulation Game; Nursing education; central venous catheter care

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either a virtual simulation game-based education group or a comparison group receiving standard education, and outcomes are assessed in parallel.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (Active Comparator): Participants in this group receive standard theoretical education on central venous catheter care management delivered through lectures and routine instructional materials as part of the nursing curriculum. No virtual simulation game is used in this group.
  Interventions: Other: Standard Nursing Education
- Virtual Simulation Game Group (Experimental): Participants in this group receive game-based virtual simulation training on central venous catheter care management.
  Interventions: Other: Virtual Simulation Game-Based Education

INTERVENTIONS:
Other: Virtual Simulation Game-Based Education — A structured virtual simulation game designed to teach evidence-based central venous catheter care management to nursing students, including interactive scenarios, clinical decision-making tasks, and immediate feedback.
  Arms: Virtual Simulation Game Group
Other: Standard Nursing Education — Classroom-based theoretical training on central venous catheter care management, routinely provided in the nursing curriculum.
  Arms: No Intervention

SUMMARY:
This study aims to evaluate the effect of virtual simulation games on developing nursing students' knowledge, skills, confidence, and satisfaction levels regarding central venous catheter care and management. Nursing students will be included in the study, and participants will take part in a virtual simulation game-based training programme. Students' knowledge levels, clinical skills, confidence, and satisfaction with the training will be assessed before and after the training using valid measurement tools. The results obtained aim to reveal whether virtual simulation games are an effective and safe teaching method in nursing education. The results of this study are expected to contribute to the development of innovative teaching methods in nursing education.

DETAILED DESCRIPTION:
This study is a planned randomised controlled trial designed to evaluate the effect of virtual simulation game-based training on developing knowledge, clinical skills, confidence, and satisfaction levels regarding central venous catheter (CVC) care and management among nursing students. The study will be conducted with students enrolled in the university's nursing programme.

Participants will be included in a structured training programme using a virtual simulation game. The training content includes evidence-based practices in central venous catheter care, infection prevention approaches, and safe care steps. The virtual simulation game is designed to allow students to experience clinical decision-making, application sequence, and error awareness in a safe learning environment.

The data collection process in the study will be carried out in two stages: pre-training and post-training. Students' knowledge levels, clinical skills, self-confidence, and satisfaction with the training will be assessed using valid and reliable measurement tools. All assessments will be conducted to determine the effect of the intervention on learning outcomes.

It is anticipated that the findings from this study will provide evidence for the use of virtual simulation games as an effective teaching method in nursing education and contribute to enhancing student competence in central venous catheter care.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the Fundamentals of Nursing course
* Must volunteer to participate in the research.

Exclusion Criteria:

* Having graduated from high school, college or university in a health-related field,
* Having taken the fundamentals of nursing course
* Having difficulty understanding and speaking Turkish.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-03-19 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Central Venous Catheter Care Management Knowledge Level | Before training (at the outset) and immediately after training is completed
  The level of knowledge of nursing students regarding central venous catheter care management will be measured using a knowledge assessment test developed based on evidence-based guidelines and validated for validity and reliability. The measurement will be conducted comparatively before and after the training. Data will be analyzed using SPSS version 26.0. Descriptive statistics will be presented as frequencies and percentages for categorical variables and as mean ± standard deviation or median (minimum-maximum) for continuous variables, as appropriate. Normality will be assessed using skewness and kurtosis values. Baseline comparability between the intervention and control groups will be evaluated using the chi-square test. Changes in knowledge, skill performance, self-confidence, and satisfaction scores before and after the intervention will be analyzed using mixed-design two-way ANOVA, with additional within- and between-group comparisons conducted using appropriate parametric or n

SECONDARY OUTCOMES:
Clinical Skill Level for Central Venous Catheter Care | Immediately after the training is completed
  The clinical skill level of nursing students regarding central venous catheter care will be assessed using a structured skills checklist. The assessment will be conducted during the post-training period.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kandemir Özsoy, Study Director — Ankara University
Locations (1):
- Ankara University Kızılcahamam Vocational School of Health Services, Kızılcahamam/ANKARA, Ankara, Kizilcahamam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data obtained in this study, with all identifying information removed, will be shared after the publication of the article, upon reasonable request and with the approval of the ethics committee, solely for the purpose of scientific research. Data sharing will take place following the signing of a data usage agreement and the evaluation of the relevant research proposal.